CLINICAL TRIAL: NCT05360836
Title: The Effect of Motor Imagery on Pain, Kinesiophobia, Functionality and Quality of Life in Patients With Radius Distal End Fracture
Brief Title: The Effect of Motor Imagery in Patients With Radius Distal End Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Melike Gizem KALAYCI, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUniversityCerrahpasa
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Distal Radius Fracture
Keywords: Fracture; Motor imagery; telerehabilitation; radius
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative (Experimental): Conservative Treatment Program
  Interventions: Other: Conservative treatment via telerehabilitation
- Motor Imagery (Experimental): Conservative Treatment + Motor Imagery Program
  Interventions: Other: Conservative treatment via telerehabilitation; Other: Conservative treatmen + motor imagery

INTERVENTIONS:
Other: Conservative treatment via telerehabilitation — Patients will do their exercises in the form of a WhatsApp video call or a Zoom video call.
  Contrast bath, massage application for 5 minutes, passive, active assistive normal range of motion. Ice application. After 4 weeks strenghtening exercise. The treatment time 8 weeks.
Other: Conservative treatmen + motor imagery — Patients will do their exercises in the form of a WhatsApp video call or a Zoom video call.
  Contrast bath, 5-minute massage, passive, active auxiliary normal range of motion. Ice application. Strengthening exercise after 4 weeks. The duration of treatment is 8 weeks. This group applies motor images for a maximum of 5 minutes. They will implement functionality-based motor images.
  Arms: Motor Imagery

SUMMARY:
Distal Radius End Fracture (DRC) is one of the most common fractures among all extremity fractures and wrist fractures . Pain, edema and functional loss are common findings in patients, and the physiotherapy program should be well planned from an early time. However, although there are different physiotherapy and rehabilitation applications in the treatment of DRC, there is not enough information about the effectiveness of the applications when the evidence-based studies are examined.

The aim of this study is to investigate the effect of motor imagery added to conventional treatment versus conventional treatment with telerehabilitation in patients with distal radius end fracture. Motor imagery is defined as the mental presentation of voluntary movement without body movement. It is an application that does not require cost and it is a training that can be easily applied in rehabilitation programs. Telerehabilitation is important in the management of patients in the acute phase of the disease, as well as in the remote management of individuals with chronic health problems. Cases who applied to Istanbul University-Cerrahpaşa Medical Faculty Orthopedics and Traumatology Clinic and were referred to Istanbul University-Cerrahpaşa Physiotherapy and Rehabilitation Department will be included in the study. Few studies have examined the effects of motor imagery on pain, kinesiophobia, and functionality in musculoskeletal injuries. Studies on the effects of motor imagery on different patient groups are needed. Therefore, in our study, the effect of motor imagery training applied with the telerehabilitation method on pain, kinesiophobia and functionality in patients with distal radius end fracture will be examined.

Sociodemographic data form of all subjects who volunteered to participate in the study; Age, gender, height, weight, pain, dominant extremity, and the type of fracture will be questioned. In addition, pain intensity is measured with a visual analog scale, normal joint movement measurement (wrist flexion, extension, ulnar and radial deviation, and forearm supination and pronation) with goniometer, hand grip strength with "Hydraulic hand dynamometer" , finger grip strength "Hydraulic Finger Dynamometer", kinesiophobia Tampa Kinesiophobia Scale, functionality "Arm, Shoulder and Hand Injury Questionnaire in Turkish (Disabilities of Arm, Shoulder and Hand-Turkish - DASH-T and The Patient-Based Wrist Assessment Questionnaire (HBEBD), with the fine dexterity Moberg Pick Up test, the motor imagery ability with the Recognize™ phone app and the Kinesthetic and Visual Imagery Questionnaire, quality of life will be evaluated with SF-12.

After the initial evaluation, the treatment program was started. Advances in the treatment method specific to the groups they belong to are explained in detail below.

Treatment:

After the distal radius end fracture, after 6 weeks of plaster application, after the first evaluation to be made in the clinic after the plaster was removed, in the next session, after patient education, conventional treatment was applied to the cases in Group 1, 3 days a week as stated below.

Group 2: Conservative Treatment + Motor Imagery Program Patients in this group will have motor imagery in addition to conservative treatment. The patients in this group will first be given a motor imagery introductory session. According to the results of the observation and evaluation made by the physiotherapist before the treatment, the function of the patients

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture and conservative treatment was decided

Exclusion Criteria:

* Bilateral fracture
* Cases with unstable, comminuted or complicated fractures, fractures associated with malignant conditions, presence of infection, cognitive impairment or inability to perceive verbal commands, and bilateral fractures will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Muscle Strenght | 3 minutes
  A dynamometer was used to evaluate muscle strength. Muscle strength was evaluated in the following muscles, each measurement was made three times and the maximum was taken.
Functionality Level | 10 minutes
  Dash, The Patient-Based Wrist Assessment Questionnaire (HBEBD)
Kinesiofobia Level | 10 minutes
  Kinesiophobia, defined as an excessive, irrational, and debilitating fear of physical movement and activity resulting from a feeling of vulnerability due to painful injury or reinjury" is found to be a central factor in the process of pain developing from acute to chronic stages .Tampa scale
Pain Level | 1 minutes
  Purpose and application of the test: The Visual Analog Scale (VAS) is used to convert some values that cannot be measured numerically into numericals. Two end definitions of the parameter to be evaluated are written on both ends of a 100 mm line and the patient is asked to indicate where his condition is appropriate by drawing a line or by placing a point or pointing on this line. Rest, activity and night were evaluated in three different time periods

SECONDARY OUTCOMES:
Normal Range of Motion | 5 minutes
  Upper extremity joints and range of motion were evaluated
the Recognize™ | 10 minutes
  Use the Recognise App to quickly exercise your synapses on your device, wherever you are.
SF-12 | From the start of treatment until 8 week after the end of treatment
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
the Kinesthetic and Visual Imagery Questionnaire | 10 minutes
  The KVIQ assesses on a five-point ordinal scale the clarity of the image (visual: V subscale) and the intensity of the sensations (kinesthetic: K subscale) that the subjects are able to imagine from the first-person perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Melike Gizem Kalaycı, PhD, Study Director — Bahçeşehir University
Locations (1):
- Melike Gizem Kalaycı, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kalayci MG, Analay Akbaba Y, Guven MF. The effect of motor imagery on functionality, pain, kinesiophobia, and quality of life in patients with distal radius fractures: A randomized controlled double-blind study. J Hand Ther. 2025 Oct-Dec;38(4):726-735. doi: 10.1016/j.jht.2025.02.018. Epub 2025 Apr 25. PMID 40287381